CLINICAL TRIAL: NCT04150523
Title: Perspectives on Prophylactic Antibiotic Use in Dermatologic Surgery: a Prospective Multi-center Cohort Study
Brief Title: Perspectives on Prophylactic Antibiotic Use in Dermatologic Surgery
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 833873
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — The study will involve a 22 question online survey, administered through the online survey platform conjoint.ly. Conjoint.ly is a web-based survey tool used to conduct survey research, evaluations and other data collection activities. Participants will complete a conjoint.ly survey and choose between treatment (antibiotic vs no antibiotic) scenarios.

SUMMARY:
This is a prospective, multi-center observational survey study to uncover how antibiotic differences can influence utilization decisions. The purpose is to assess the trade-offs between drug side effects and infection prevention that patients are willing to make when taking prophylactic antibiotics. Misuse of antibiotics or non-adherence to prescribed regimens is a public health issue that may be due to a variety of reasons including unclear instructions, symptom improvement and adverse events Subjects will be healthcare providers (physician or nurse) and individuals 18+ years of age in the dermatologic surgery waiting area (including patients and accompanying individuals). Participants will complete a conjoint.ly survey and choose between treatment (antibiotic vs no antibiotic) scenarios.

DETAILED DESCRIPTION:
This is a prospective, multi-center observational survey study to uncover how antibiotic differences can influence utilization decisions. The purpose is to assess the trade-offs between drug side effects and infection prevention that patients are willing to make when taking prophylactic antibiotics. Misuse of antibiotics or non-adherence to prescribed regimens is a public health issue that may be due to a variety of reasons including unclear instructions, symptom improvement and adverse events Subjects will be healthcare providers (physician or nurse) and individuals 18+ years of age in the dermatologic surgery waiting area (including patients and accompanying individuals). Participants will complete a conjoint.ly survey and choose between treatment (antibiotic vs no antibiotic) scenarios.

Adults in the dermatologic surgery department waiting room with age greater than or equal to 18 years (this includes both patients and accompanying individuals (family members, friends, caregivers)) and healthcare providers in dermatologic surgery. A member of the study team will approach patients in the Perelman Dermatology Clinic to determine if they meet inclusion criteria and educate them about the study using the verbal script. If interested, patients will receive a link to the online survey, which will contain an informed consent page. Dermatology healthcare providers will be identified in clinic or from academic center staff directories. Individuals meeting inclusion criteria will also be recruited from the dermatologic surgery waiting rooms of other collaborating institutions (Penn State Health, University of Missouri Health Care, Indiana University Health, University of Minnesota, Oregon Health & Science University, Washington University in St. Louis, UT Southwestern, UC Davis and Ohio State University) once approved by their IRB.

All data will be collected and stored in a secured password-protected conjoint.ly account managed by the Penn Dermatologic Surgery Clinical Research Team. Collaborating institutions will not have access to the survey responses. Data analysis: Multivariate random parameters logit will be used to estimate preference weights for each attribute level. These preference weights will be used to estimate the maximum acceptable risk of various side effects that subjects would be willing to accept in exchange for infection prevention. Collaborating researchers from other institutions will not be involved in data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Individual in the dermatologic surgery waiting room: patient, caregiver, family member or accompanying individual to patient receiving dermatologic surgery service, or dermatology healthcare provider

Exclusion Criteria:

* Age less than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults in the dermatologic surgery department waiting room with age greater than or equal to 18 years (this includes both patients and accompanying individuals (family members, friends, caregivers)) and healthcare providers in dermatologic surgery. A member of the study team will approach patients in the Perelman Dermatology Clinic to determine if they meet inclusion criteria and educate them about the study using the verbal script. If interested, patients will receive a link to the online survey, which will contain an informed consent page. Dermatology healthcare providers will be identified in clinic or from academic center staff directories.
Sampling Method: Non-Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Trade-offs | Oct 3 2019-July 1 2021
  Determine the trade-offs between surgical site infection prophylaxis and antibiotic-associated adverse effects that patients, healthcare providers and caregivers are willing to make

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California, Davis, Davis, California
  - Indiana University, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri Health Care, Columbia, Missouri
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bae-Harboe YS, Liang CA. Perioperative antibiotic use of dermatologic surgeons in 2012. Dermatol Surg. 2013 Nov;39(11):1592-601. doi: 10.1111/dsu.12272. Epub 2013 Jul 18. PMID 23865410
- [Background] Barbieri JS, Bhate K, Hartnett KP, Fleming-Dutra KE, Margolis DJ. Trends in Oral Antibiotic Prescription in Dermatology, 2008 to 2016. JAMA Dermatol. 2019 Mar 1;155(3):290-297. doi: 10.1001/jamadermatol.2018.4944. PMID 30649187
- [Background] Barbieri JS, Etzkorn JR, Margolis DJ. Use of Antibiotics for Dermatologic Procedures From 2008 to 2016. JAMA Dermatol. 2019 Apr 1;155(4):465-470. doi: 10.1001/jamadermatol.2019.0152. PMID 30825412
- [Background] Pechere JC. Parameters important in short antibiotic courses. J Int Med Res. 2000;28 Suppl 1:3A-12A. PMID 11092225
- [Background] Pechere JC. Patients' interviews and misuse of antibiotics. Clin Infect Dis. 2001 Sep 15;33 Suppl 3:S170-3. doi: 10.1086/321844. PMID 11524715
- [Background] Sclar DA, Tartaglione TA, Fine MJ. Overview of issues related to medical compliance with implications for the outpatient management of infectious diseases. Infect Agents Dis. 1994 Oct;3(5):266-73. PMID 7866659